CLINICAL TRIAL: NCT04081207
Title: A Preliminary Study of the Neurobiology of AAC-Induced Language Recovery in Post-Stroke Aphasia
Brief Title: Using Augmentative & Alternative Communication to Promote Language Recovery for People With Post-Stroke Aphasia
Acronym: NAIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Aimee Dietz, Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R15DC017280-01 (NIH)
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Post-stroke Aphasia; Aphasia
Keywords: augmentative and alternative communication; aphasia; fMRI; DTI; neuroimaging
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Intervention Model Description: Participant cohorts: We will use a 2 (groups) X 4 (measurement time points) switching replications design[18] to examine the effects of AAC on aphasia severity and spoken language (AIM 1), elucidate the neurobiological mechanism of AAC-induced language recovery (AIM 2), and identify AAC treatment responder subgroups (Exploratory Aim). This design will allow Group 2 to serve as the control group; however, they will still receive AAC treatment; thus, allowing us to increase the total N who receives AAC treatment to 20 people.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AAC-LaRc (Experimental): all participants receive the experimental treatment
  Interventions: Behavioral: AAC for Language Recovery (AAC-LaRc)

INTERVENTIONS:
Behavioral: AAC for Language Recovery (AAC-LaRc) — iPads will be programmed with a personalized communication application (app) and a structured 4-step intervention will be employed to instruct patients how to cue themselves during anomic events via pictures, text, or speak buttons.

SUMMARY:
The currently available interventions only partially restore language abilities in patients with post-stroke aphasia; preventing successful reintegration into society. This study will increase our knowledge of how we can use assistive technology interventions to help people with aphasia restore language function. Further, this project will help us identify regions of the brain responsible for these changes.

DETAILED DESCRIPTION:
In aphasia rehabilitation, usual care is focused on helping people recuperate as much of their pre-stroke language capacity as possible.Typically, usual care is a non-standardized therapy that is tailored to the specific needs of the person with aphasia.Once a person reaches a plateau in language recovery, AAC is implemented with a focus on circumventing, or compensating for the communication challenges associated with aphasia.

The ability of people with aphasia to (1) recover language function well-into the chronic phase of stroke recovery and (2) self-cue to promote word retrieval during anomic events offer the solution for how AAC could be employed as a dual-purpose tool to augment language recovery and compensate for deficits. This approach, however, this requires a shift in how AAC is implemented. With the goal of language recovery, treatment needs to focus on instructing people with aphasia how to use AAC as a mechanism for self-cueing, rather than as a tool to replace speaking. Based on our pilot data, we hypothesize that this novel method to AAC implementation will promote language recovery by coupling the canonical language and visual processing neural networks.

This work will also contribute to our ability to identify, a priori, who will respond to this particular AAC intervention and who will not, by combining neuroimaging with behavioral and clinical data. This has the potential to reduce the cost of healthcare for stroke recovery by implementing the most effective treatment possible. Importantly, when we identify non-responders, this will allow us to construct a profile and identify features of the AAC treatment that require adjustment to meet their unique needs.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* native speaker of american English
* compatible for 3 Tesla MRI
* Ischemic, left middle cerebral artery stroke
* at least 12 months post stroke
* pass hearing screening
* pass vision screening
* diagnosis of aphasia on the Western Aphasia Bedside Screen
* ability to produce 5-10 intelligible words
* no more than a moderate apraxia of speech or dysarthria
* minimal or no AAC/iPad experience
* written consent by self or guardian

Exclusion Criteria:

* fails to meet the above
* Underlying degenerative or metabolic disorder or supervening medical illness
* Severe depression or other psychiatric disorder
* Report of pregnancy by women of childbearing age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Western Aphasia Battery-Revised Aphasia Quotient | 3 years
  a diagnostic tool used to determine aphasia type and severity
Visual Regions of Interest Activation intensity | 3 years
  A functional magnetic resonance imaging (fMRI) measure to indicate change in brain involvement during resting state and language tasks.
Connectivity Indices | 3 years
  Connectivity indices reflect the temporal correlation between canonical language and visual regions of interest during language and resting state fMRI tasks.

SECONDARY OUTCOMES:
Motor-Free Visual Perception Test-4 | 3 years
  The Motor-Free Visual Perception Test-4 assesses visual perceptual ability without requiring motor responses.
Discourse Analyses | 3years
  We will calculate percentage of counted words, mazes, correct information units, t-units, during personal story retells with and without the AAC support.
Communication analyses | 3 years
  We will calculate percentage of communication conveyed via pictures, text boxes, and speak button during personal story retells with and without the iPad AAC support.
Stroke and Aphasia Quality of Life-39 (SAQOL-39) | 3 years
  The SAQOL-39 is a valid and reliable measure of health related quality of life, post-stroke that uses an aphasia friendly 5 point Likert scale format.
Communication Effectiveness Index (CETI) | 3 years
  The CETI measures functional communication scenarios that caregivers rate the ability of the patient to complete tasks, as compared to before their stroke, via a 10 cm visual analogue scale.
Fractional Anisotropy (FA) | 3 years
  FA is a value of diffusion and reflects white matter density and myelination. We will examine the following tracts: (1) superior, (2) inferior fronto-occipital, (3) middle longitudinal, (4) inferior longitudinal fasciculus, (5) arcuate, and (6) uncinate
Mean Diffusivity (MD) | 3 years
  MD is used to map tracts and serves as a measure of health or disease in white matter. We will determine the MD for the following pathways: (1) superior, (2) inferior fronto-occipital, (3) middle longitudinal, (4) inferior longitudinal fasciculus, (5) arcuate, and (6) uncinate
Language Lateralization Indices (LI) | 3 years
  LI is a measure that reflects hemispheric dominance for language, while accounting for lesioned tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Dietz, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Even though the final dataset will be stripped of identifiers prior to release for sharing, we believe that there remains the possibility of deductive disclosure of subjects based on their private health information and language profiles. Further, it is possible to reconstruct faces from MRI data and the patients are easily identified through the testing and treatment videos; thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. Data will be shared at the time of publication, or shortly thereafter.
Supporting Information: Study Protocol, ICF
Time Frame: Upon study completion

REFERENCES:
- [Background] Dietz A, Vannest J, Maloney T, Altaye M, Holland S, Szaflarski JP. The feasibility of improving discourse in people with aphasia through AAC: Clinical and functional MRI correlates. Aphasiology. 2018;32(6):693-719. doi: 10.1080/02687038.2018.1447641. Epub 2018 Mar 9. PMID 32999522